CLINICAL TRIAL: NCT05031364
Title: Effectiveness of Evidence-Based Mental Health Practices for Youth With Autism Supported by Online Consultation to Practitioners in Community and Navy Clinics
Brief Title: CBT for Youth With Autism and Emotional/Behavioral Needs in Community Care Settings
Acronym: CYAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Virginia Commonwealth University (Other); United States Naval Medical Center, San Diego (U.S. Federal Agency); Westside Regional Center (Unknown); California Autism Professional Training and Information Network (Unknown)
Responsible Party: Principal Investigator, Jeffrey J. Wood, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AR200108
Record Dates: First submitted 2021-07-28; First posted 2021-09-01 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Treatment condition and timepoint will be masked for the outcomes assessors (independent evaluators [IEs]), who will administer the interview-based measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consultation-Based Training on BIACA (Experimental): Community mental health clinicians will be given online one-on-one training and consultation in the BIACA (Behavioral Interventions for Anxiety in Children with Autism; e.g., Wood et al., 2020) CBT program. Clinicians will be provided with weekly 30-minute video-conference-based consultation sessions with an expert in BIACA. These consultation sessions are manual-driven and utilize a Practice-Based Coaching format, in which a trained consultant meets weekly with clinicians to provide practice-based feedback (cf. McLeod et al., 2018). Consultation meetings include agenda setting, case material review, planning for the next treatment session, and a meeting summary. Relevant online training materials (e.g., demonstration videos of CBT sessions; corresponding written session materials) developed in the context of a NIMH R34 grant available on meya.ucla.edu (1R34MH110591) will also be provided to clinicians for each upcoming therapy session.
  Interventions: Behavioral: Behavioral Interventions for Anxiety in Children with Autism (BIACA)
- Usual Care Augmented by Self-Instruction Resources for CBT for Autism (Active Comparator): Community mental health clinicians in this arm will provide any therapy, counseling, and/or behavioral treatment procedures they deem appropriate for each participating child. Clinicians randomized to this arm will be given immediate access to CBT-for-autism self-instruction materials that are already freely available to any clinician at meya.ucla.edu (see Consultation-Based Training on BIACA arm, above), to supplement their usual clinical care, if they so choose, until they complete their Usual Care/Self-Instruction participation and are offered direct training and weekly consultation in BIACA.
  Interventions: Behavioral: Treatment-as-Usual Supplemented by Internet-Based Self-Instruction (MEYA)

INTERVENTIONS:
Behavioral: Behavioral Interventions for Anxiety in Children with Autism (BIACA) — In the BIACA CBT program (e.g., Wood et al., 2020), clinicians work with families for 16 weekly sessions that include both the child and parent(s). In BIACA, anxiety, rigidity and inflexible routines, and irritability are all addressed using in vivo exposure therapy strategies during sessions as well as parent (and teacher) training to promote regulation across settings. ASD-related clinical needs that can impact mental health and emotion regulation such as friendship skills and social entry skills (e.g., joining games at school) are addressed with modeling, self-management, and parent- (or teacher-) implemented social coaching in daily settings. For youth with limited communication, therapy is adapted through the use of play-based representations of challenging situations and an emphasis on more action-oriented exposure therapy.
  Arms: Consultation-Based Training on BIACA
Behavioral: Treatment-as-Usual Supplemented by Internet-Based Self-Instruction (MEYA) — Participating clinicians are expected to have varied training in numerous psychological therapy procedures (e.g., insight-oriented procedures, cognitive interventions, family therapy, etc.), any or all of which they may choose to implement with a participating child. These practices will be characterized through the Therapy Procedures Checklist (Weersing et al., 2002). Additionally, participating clinicians will be provided with information about self-instruction resources on CBT for children with autism, namely, the Modular Evidence-Based Practices for Youth with Autism (MEYA) website developed by our research group. MEYA is freely accessible to clinicians worldwide at meya.ucla.edu. MEYA incorporates treatment elements of both BIACA (Wood et al., 2020) and SEBASTIEN (Wood et al., 2021), which was designed to address additional autism-related clinical needs (e.g., reciprocal conversation). Clinicians in this arm will provide up to 16 therapy sessions.
  Arms: Usual Care Augmented by Self-Instruction Resources for CBT for Autism

SUMMARY:
This study is a 4-year randomized, controlled trial comparing cognitive behavioral therapy (CBT) to usual clinical care for children (aged 6-14 years) with autism and emotional dysregulation (e.g., irritability, anxiety). We will randomly assign 50 mental health clinicians, each treating 2 youth (N = 100 youth total), to CBT program for emotional dysregulation and core autism symptoms with weekly live consultation with an expert or to usual clinical care augmented by self-instruction in CBT, in a 1:1 allocation. The CBT manual is well-supported in our efficacy research, has been replicated in other centers, is free/open-access (meya.ucla.edu), and has user-friendly digital and traditional print materials for mental health clinicians (e.g., psychologists, counselors) to use in preparing for and conducting therapy sessions. The primary outcome measure will be assessed weekly. Additional assessments will occur at Screening, Mid-treatment, Post- treatment and 3-month Follow-up.

ELIGIBILITY:
Clinician's inclusion criteria: All practitioner participants will regularly treat at least some youth with ASD within a recognized field of practice (e.g., clinical psychology, counseling, marital and family therapy, social work) and will serve youth with ASD referred by the Regional Centers, Tricare/NMCSD, or the California public schools. Practitioners will agree to invite one or more potentially eligible families of youth with ASD so that, in total, at least 2 of the new families referred to them participate in the study (i.e., each clinician will aim to have a cluster of two families randomized to the same condition with them; however, the two referrals can be non-parallel and clinicians will not be required to enroll a second client to remain in the study, since there is no way for them to guarantee future enrollment from client families. As needed, additional clinicians can be enrolled in the study to reach the target of 100 youth.). Up to four families per practitioner will be allowed so long as the minimum study enrollment of at least 50 practitioners and 100 client families randomized is met.

Youth inclusion criteria: Youth participants will be boys or girls between 6 and 14 years of age with a documented clinical diagnosis of ASD and will be newly referred for outpatient services with a participating clinician. Additional eligibility criteria are as follows:

1. Youth will have a pre-existing clinical diagnosis of ASD made by an appropriate licensed professional (e.g., clinical psychologist, developmental pediatrician) which will be documented in a report or medical note provided by the family, or confirmed telephonically by the diagnosing professional.
2. The parent-reported Social Responsive Scale-2 (SRS-2; Constantino & Gruber, 2012) Total T-Score will be > 60 (cut-score maximizing ROC curve parameters for screening for ASD; area under the curve = 98.8%; Schanding et al., 2011).
3. Youth will meet criteria for clinically significant emotion dysregulation symptoms as defined by a minimum T-score of 60 on the Externalizing or Internalizing subscales of the parent-reported Brief Problem Monitor (BPM) and at least 15 T-score points over 50 between these two BPM subscales (e.g., Internalizing=60 + Externalizing=55).
4. The youth has a Vineland Adaptive Behavior Scales-3 Communication Composite Standard Score > 60 and Expressive Communication subscale v-score > 8 (in both cases > 1st %ile).

Exclusion Criteria:

1. For participants presenting with severe comorbid symptomology (e.g., psychotic symptoms), the comorbid conditions cannot be sufficiently severe to warrant immediate treatment or require ongoing medication titration.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Brief Problem Monitor (BPM) | Baseline (week 0), Sessions 1 to 16 (weekly, approximately weeks 1 to 16), and Follow-up (approx. week 29)
  The BPM (Achenbach et al., 2011) is an abbreviated version of the widely used Child Behavior Checklist (CBCL; Achenbach & Rescorla, 2001). The sum of the parent-report BPM Internalizing and Externalizing subscales will be utilized as the primary outcome measure in this study to index improvement across core aspects of children's mental health (i.e., anxiety, irritability, depressed mood, defiance). The BPM is comprised of 19 items. Each item is rated 0 = not true, 1 = somewhat true, or 2 = very true. Higher scores reflect more problems. Research suggests the BPM has good reliability and validity and is sensitive to change in effectiveness studies of youth psychotherapy (Piper et al., 2014; Weisz et al., 2012). The BPM can be administered remotely via the internet.

SECONDARY OUTCOMES:
Change in Youth Top Problems (YTP) Rating Scale | Baseline (week 0), Sessions 1 to 16 (weekly, approximately weeks 1 to 16), and Follow-up (approx. week 29)
  The YTP approach is a valid and reliable personalized assessment method that is sensitive to psychotherapy treatment response in children that allows clinicians and researchers to identify problems of the children or adolescents that are especially important from the perspective of a caregiver (Weisz et al., 2011,2012). The YTP caregiver interview (YTP-P) will be administered after Vineland and SACA at screening. This interview allows caregivers to state in their own words what "current" symptoms/problems experienced by their child are the most concerning to them. The specific problems are transcribed in the parents' own words. Interviewers then obtain Initial YTP Symptom Severity Ratings for each problem on a scale ranging from 0 (not at all) to 10 (very, very much). The top 12 problems will then be rated weekly throughout the child's therapy by the caregiver. Higher scores reflect more significant problems.
Change in Social Responsiveness Scale II (SRS-II) | Baseline (week 0), Session 8 (approximately week 8), Immediate Post-Treatment [approx. week 16], and Follow-up (approx. week 29)
  The SRS-II (Constantino & Gruber, 2012) is a 65-item parent-rated scale measuring the severity of ASD symptoms. The SRS-II has high internal consistency, convergence with other measures of ASD severity, and discriminates between youth with and without ASD (Schanding et al., 2011). It has shown treatment sensitivity in all extant clinical trials of BIACA including the replications by Storch and colleagues; versus treatment-as-usual; and versus standard-of-practice CBT (e.g., Storch et al., 2013, 2015; Wood et al., 2009b, 2015a, 2020).
Consumer Satisfaction Parent Questionnaire | Immediate Post-Treatment [approximately week 16]
  Parent satisfaction with treatment will be assessed with an 11-item parent-report measure.

OTHER OUTCOMES:
Therapy Procedures Checklist (TPC) | Immediate Post-Treatment [approximately week 16]
  The TPC (Weersing et al., 2002) is a 62-item self-report measure used to assess practitioners' use of treatment techniques that correspond to cognitive, behavioral, psychodynamic, or family orientations. Techniques in each orientation are summed to create total scores, with higher scores reflecting more extensive use of techniques consistent with that orientation. The TPC has excellent internal consistency and test-retest reliability (Baumann et al., 2006; Weersing et al., 2002). Item scores range from 1 (rarely) to 5 (most of the time).
The Modular EBPs for Youth with Autism Fidelity Scale (MEYA-FS; McLeod et al., 2022) | Sessions 1 [approximately week 1], 5 [approx. week 5], 9 [approx. week 9], and 13 [approx. week 13]
  The MEYA-FS is a 32-item measure designed to assess clinician adherence and competence for practices found in EBPs for autistic youth. Beginning in session 1, and then every 4 sessions thereafter, clinicians in both treatment arms will record their treatment session with the child and family. These recordings will be rated by trained IEs using the BIACA Fidelity Scales. Coders are asked to estimate the extent to which clinicians engage in each strategy during a session using a 7-point Likert-type scale with the following anchors: 1=not at all, 3=somewhat, 5=considerably, 7=extensively. Higher scores reflect greater adherence and competence.
Change in BIACA Therapist Quiz | Baseline [week 0] and Immediate Post-Treatment [approximately week 16]
  The BIACA Therapist Quiz assesses clinicians' knowledge of BIACA concepts and clinical scenarios. This measure will be administered to clinicians at pretreatment and posttreatment to assess development of CBT knowledge through the process of training and consultation in BIACA.
Mixed-methods feedback on training and consultation in BIACA | Immediate Post-Treatment [approximately week 16]
  Acceptability and feasibility of training/consultation in BIACA will be assessed quantitatively using the Evidence-Based Practice Attitude Scale (Aarons, 2004) and the Usage Rating Profile-Intervention (Chafouleas et al., 2011). We will review answers on the measures and use them to guide approximately 20-minute semi-structured interviews with the mental health clinician at the end of the acute treatment for clinicians in the BIACA arm. In addition, the following areas will be queried in these interviews: the quality and strengths/weaknesses of the online training and consultation interface (e.g., length and content of training and session materials and videochat consultations), system efficiency (how much time was put into the weekly session preparation and was this viewed as too much or acceptable), and clinical strategies as applied to their clients. Recorded interview responses will be transcribed.

CONTACTS AND LOCATIONS:
Overall Officials: Wood, Principal Investigator — University of California
Locations (3):
- United States (3):
  - Westside Regional Center, Culver City, California
  - California Autism Professional Training and Information Network (CAPTAIN), Sacramento, California
  - Naval Medical Center San Diego, San Diego, California

IPD SHARING:
Plan to Share IPD: Yes
To comply with the Policy, we propose to make de-identified data, codebooks, and documentation available under the auspices of the National Database for Autism Research (NDAR) (for data) and the PI's UCLA website (for codebooks, documentation, etc.). The study protocol is posted on clinicaltrials.gov.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Datasets associated with manuscripts that are published during or following the grant period will be available once each manuscript is made available by the publisher. The final data set will be made available from Dr. Wood within 3 years after the end of all data collection activities. All datasets will be stored and made available for a minimum of 10 years or longer, depending on the extant NDAR policies.
Access Criteria: NDAR sets a universal policy for accessing its datasets. Other information will be freely available on the PI's website.

REFERENCES:
- [Background] Wood JJ, Kendall PC, Wood KS, Kerns CM, Seltzer M, Small BJ, Lewin AB, Storch EA. Cognitive Behavioral Treatments for Anxiety in Children With Autism Spectrum Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2020 May 1;77(5):474-483. doi: 10.1001/jamapsychiatry.2019.4160. PMID 31755906
- [Background] Wood JJ, Ehrenreich-May J, Alessandri M, Fujii C, Renno P, Laugeson E, Piacentini JC, De Nadai AS, Arnold E, Lewin AB, Murphy TK, Storch EA. Cognitive behavioral therapy for early adolescents with autism spectrum disorders and clinical anxiety: a randomized, controlled trial. Behav Ther. 2015 Jan;46(1):7-19. doi: 10.1016/j.beth.2014.01.002. Epub 2014 Jan 22. PMID 25526831
- [Background] Wood JJ, McLeod BD, Klebanoff S, Brookman-Frazee L. Toward the implementation of evidence-based interventions for youth with autism spectrum disorders in schools and community agencies. Behav Ther. 2015 Jan;46(1):83-95. doi: 10.1016/j.beth.2014.07.003. Epub 2014 Jul 30. PMID 25526837
- [Background] Lecavalier L, Wood JJ, Halladay AK, Jones NE, Aman MG, Cook EH, Handen BL, King BH, Pearson DA, Hallett V, Sullivan KA, Grondhuis S, Bishop SL, Horrigan JP, Dawson G, Scahill L. Measuring anxiety as a treatment endpoint in youth with autism spectrum disorder. J Autism Dev Disord. 2014 May;44(5):1128-43. doi: 10.1007/s10803-013-1974-9. PMID 24158679
- See also: Online repository of CBT practices used in the training/consultation protocol. — http://meya.ucla.edu

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-30): https://cdn.clinicaltrials.gov/large-docs/64/NCT05031364/Prot_SAP_000.pdf